CLINICAL TRIAL: NCT05682508
Title: Efficiency of Education Based on Health Belief Model in Diet and Fluid Control of Hemodialysis Patients
Brief Title: Effect of Educution in Control Nutrition and Fluid Control of Hemodialysis Patient
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ufuk DEMİREL, Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/15
Record Dates: First submitted 2023-01-01; First posted 2023-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-01

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; education; Health Belief Model; nursing
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant: Patients in the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education group (Experimental): The training planned four step. In the first interview, a pre-test will be applied by the researcher. The patient will then be trained and given a training booklet. The second interview will take place 30 days after the end of the first training. The topics will be summarised and the benefits of adherence to diet and fluid control will be emphasised. The third interview will be held 30 days after the second interview. In this interview, the patient's questions will be answered and the necessary training sections will be explained again for patient. The issues that prevent the patient from complying with fluid and diet control will be discussed with the patient and positive developments in the patient prognosis will be reinforced. The last interview will be held 30 days after the third interview. In all interviews, data will be collected with data collection tools and clinical parameters of the patient will be recorded.
  Interventions: Other: Education group
- Control grup (No Intervention): No training will be given to the control group. In the first interview will be applied data collection tools and will be recorded clinical parameters. Last interview with control group will be held 90 days after first interview. Data collection tools will be applied and clinical parameters will be recorded in last interview. The training booklet will be given also to patients in control group at the end of the research.

INTERVENTIONS:
Other: Education group — Based on the Health Belief Model, a "educational booklet on diet and fluid control in individuals receiving hemodialysis treatment" has been prepared. The training content consists of information on the structure and function of the kidneys, information about chronic renal failure, possible complications in case of non-adherence with the desired fluid control and diet, perceived benefits, the information on diet and fluid control consisted of perceived benefits, barriers, coping with barriers, perceived susceptibility in this regard, and information on the development of self-efficacy to improve dietary compliance and fluid control.
  Individuals in the education group were given individual training by the researcher. The training was conducted in a single meeting of 20-30 minutes in the first hour when haemodialysis started and the patient's condition was stable.
  Arms: Education group

SUMMARY:
Hemodialysis patients are required to adhere to diet and fluid restriction. The literature shows that hemodialysis patients have low adherence to diet and fluid restriction.

Failure to adhere to fluid control increases weight gain between two dialysis sessions. Increased weight gain between two dialysis sessions can lead to signs and symptoms, such as heart failure, hypertension, edema and dyspnea. Ultrafiltration is increased during dialysis to remove excess fluid from the body between two dialysis sessions. As a result, this leads to large changes in the patient's weight during dialysis sessions, leading to hemodialysis complications such as hypotension and muscle cramps.

Diet is important to prevent uremic complication for hemodialysis patient. Diet restriction purposes to minimize uremic symptoms and fluid- electrolyte imbalance. As increase failure to adhere diet, serum phosphorus serum potassium rise and weight gain between two dialysis sessions increases. As a result, problems with the cardiac system, respiratory system and bones are experienced.

Diet and fluid restriction helps to prevent complications, to increase the quality of life and to reduce mortality. Therefore, diet and fluid control vitally important for hemodialysis patients.

Nurses have an important place in providing diet and fluid management. Desired success can be achieved in fluid and diet control by giving planned trainings to patients by nurses. In patient education, the Health Belief Model is used as an effective guide, which explains the reason for the person's attitudes and behaviors. This model is based on explain why did the patient not adhere with the treatment and what motivates the patient. The model is based on the premise that they will change their behavior when people understand the severity of the illness.

The Health Belief Model can used education on diet and fluid contol of hemodialysis patients. In this study, Health Belief Model components will be used as a guide in the preparation of the educational content to be given to hemodialysis patients. With this study planned to be done; it was aimed to determine the effect of Health Belief Model-based education on diet and fluid control of hemodialysis patients. The study was planned as a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* He is over 18 years old,
* At least 6 months of hemodialysis treatment,
* At least primary school graduate,
* Does not have a condition that interferes with language, hearing or visual communication,
* Patients who accept to participate in the study are included in the study

Exclusion Criteria:

* That do not meet the inclusion criteria,
* Those who are included in another training program on the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | up to 1 year
  It was prepared by the researchers by analysing the relevant literature.
  In the personal information form, socio-demographic and disease information of the patient were questioned.

SECONDARY OUTCOMES:
Fluid Control Scale in Haemodialysis Patients | up to 1 year
  It was developed by Albayrak Coşar and Çınar (2012) to measure the knowledge, behaviours and attitudes of haemodialysis patients about fluid restriction. The scale was prepared in the form of a 3 point Likert-type scale. The participants were asked to respond to each item as "agree", "indecisive", or "don't agree". When assessing positive items, "agree" was scored 3, "indecisive" 2, and "don't agree" 1. The negative items (6, 7, and 18-24) are reversely scored. The lowest score obtained from the scale is 24 and the highest score is 72. As the score obtained from the scale increases, patients' compliance with fluid control also increases

OTHER OUTCOMES:
Dietary Knowledge Scale of Hemodialysis Patients | up to 1 year
  It was developed by Bulantekin Düzalan and Cınar Pakyuz in 2014. It was developed to evaluate the dietary knowledge of patients with ESRD receiving haemodialysis treatment. The scale consists of 18 items and is 3-point Likert type . The scoring was as follows: True: "1" point; False: "0" points; and I don't know: "0" points. The lowest and highest scores were 0 and 18 points, respectively. The scale consisted of a single sub-dimension and there was one reverse-scored item (12th item). The scale did not contain a cut-off score and the interpretation was "a good level of knowledge" for higher scores.
Scale for Dietary Behaviours in Haemodialysis Patients | up to 1 year
  It was developed by Bulantekin Düzalan and Cınar Pakyuz in 2014. The scale was developed as a five-point Likert scale with these options: "strongly disagree, disagree, not sure, agree, and strongly agree", ranging from 1 to 5 points, respectively. The scale consisted of a single sub-dimension and there were no reverse-scored items. The lowest and highest scores were 13 and 65 points, respectively. The scale did not contain a cut-off score and the interpretation was "a good behavioural status" for higher scores.
Clinical Parameter Monitoring Form | up to 1 year
  The form was prepared by the investigators to record blood pressure, interdialytic weight gain, dry weight, ultrafiltration value and biochemistry values of the patients. The data in the patient file will be used for the relevant laboratory values of the patient and no new tests will be requested.

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Demirel, Principal Investigator — Ege University
Locations (1):
- Zonguldak Atatürk Public Hospital, Zonguldak, Center, Turkey (Türkiye)